CLINICAL TRIAL: NCT02660905
Title: Evaluation of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (ECF/TAF) Switch Followed by Ledipasvir-Sofosbuvir HCV Therapy in HIV-HCV Co-Infection: A CIHR Canadian HIV Trials Network-Gilead Pilot Trial Proposal
Brief Title: HIV Drug Switch Followed by HCV Therapy in HIV-HCV Co-Infection
Acronym: CTN289
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Gilead Sciences (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150881-01H
Record Dates: First submitted 2015-10-21; First posted 2016-01-21 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2019-03

CONDITIONS: Human Immunodeficiency Virus; Hepatitis C, Chronic
Keywords: HIV-HCV co-infected; HCV; HIV; Hep C; Hepatitis C; HCV positive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic; Hepatitis C | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Rilpivirine; Tenofovir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Treatment (Experimental): E/C/F/TAF Ledipasvir-Sofosbuvir/TAF
  Interventions: Drug: E/C/F/TAF;; Drug: Ledipasvir-Sofosbuvir

INTERVENTIONS:
Drug: E/C/F/TAF; — Evaluation of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Switch followed by Ledipasvir-Sofosbuvir Antiviral HCV Therapy
  Other Names: Genvoya; emtricitabine/ rilpivirine/ tenofovir disoproxil fumarate
Drug: Ledipasvir-Sofosbuvir — Evaluation of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Switch followed by Ledipasvir-Sofosbuvir Antiviral HCV Therapy
  Other Names: Harvoni

SUMMARY:
This is an prospective open label pilot study conducted over 32 weeks.

A total of 25 eligible participants who are infected with HCV and HIV will be recruited from 2 Canadian HIV Trials Network (CTN) sites (Ottawa Hospital Research Institute and McGill University Health Centre)

This study is investigating the effectiveness of a combination of Elvitegravir/Cobicistat/Emtricitabine/ Tenofovir Alafenamide Single Tablet Regimen (E/C/F/TAF STR) for HIV treatment and Harvoni for HCV treatment.

This study will assess the effect that the study drug has on the metabolism of sugar, the changes in fat in the bloodstream, and other metabolic changes. Metabolism is the process your body uses to get or make energy from the food you eat.

This study may provide information on the impact of liver fibrosis (scarring of liver tissues) on metabolic changes before, during and after HCV antiviral therapy.

Drug-drug interactions (DDI) between E/C/F/TAF and LPV-SOF have been well evaluated and no clinically significant interactions have been identified.

A switch to E/C/F/TAF in the context of LPV-SOF HCV antiviral treatment preparation may be particularly beneficial because of its:

1. favorable side effect profile
2. once daily STR formulation
3. known DDI profile with LPV-SOF
4. neutral effect on liver fibrosis
5. improved kidney and bone safety profile with the use of TAF

Conduct of this study is justified as it:

1. Assesses a minimal pill count and dosing frequency strategy of co-treatment of HIV and HCV using well tolerated medications with an excellent safety profile and known DDI profile.
2. Provides additional safety data for TAF in the HIV-HCV co-infected population.
3. Quantifies adherence and identifies obstacles to full adherence in this population. There is a paucity of data related to DAA adherence in licensing studies.
4. Provides real-world safety and efficacy data to support the public funding for LPV-SOF DAA therapy in HIV-HCV co-infected populations.
5. Provides preliminary data on the immunologic and metabolic consequences of HCV clearance in HIV-HCV co-infection
6. As a pilot study, the information gathered will inform the feasibility of future clinical trials evaluating novel treatment strategies for HIV-HCV co-infected patients.

DETAILED DESCRIPTION:
The availability of interferon (IFN)-free HCV Direct Acting Antiviral (DAA) antiviral therapy such as Ledipasvir-Sofosbuvir (LPV-SOF) allows for broad provision of treatment for populations living with HIV-HCV. Co-infected persons frequently have competing co-morbidities and are at risk for progressive liver disease which makes adherence and combined management of HIV and HCV challenging. Simple, safe, well tolerated regimens with few drug-drug interactions could be highly beneficial in ensuring success of HCV therapy in this population. With this is mind, the optimal management of antiretroviral therapy prior to initiating LPV-SOF treatment remains unclear.

E/C/F/TAF [elvitegravir-cobicistat-emtricitabine-tenofovir alafenamide fumarate (TAF)] will be assessed in this study because it is formulated as a single tablet which facilitates adherence by once daily dosing and reduced pill count. It is established to be affective at achieving and maintaining HIV virologic suppression. The safety profile of this HIV regimen is excellent. The E/C/F/TAF formulation assessed in this study will contain TAF. This formulation has been evaluated in HIV-infected populations and found to be of equivalent HIV antiviral activity and to have improved impact on renal and bone metabolism [ref: David Wohl, Anton Pozniak, Melanie Thompson, Edwin DeJesus, Daniel Podzamczer, Jean-Michel Molina, Gordon Crofoot, Christian Callebaut, Hal Martin, Scott McCallister. Tenofovir Alafenamide (TAF) in a Single-Tablet Regimen in Initial HIV-1 Therapy. Conference on Retroviruses and Opportunistic Infections. 113LB. February 23-26, 2015, Seattle, Washington.]. There is minimal safety data in HIV-HCV co-infection.

Drug-drug interactions (DDI) between HIV antiretrovirals and HCV antivirals remain a key obstacle to the safe and effective delivery. The DDI between E/C/F/TAF and LPV-SOF have been well evaluated and no clinically significant interactions have been identified.

A switch to E/C/F/TAF in the context of LPV-SOF HCV antiviral treatment preparation may be particularly beneficial because of its:

1. favorable side effect profile
2. once daily STR formulation
3. known DDI profile with LPV-SOF
4. neutral effect on liver fibrosis
5. improved kidney and bone safety profile with the use of TAF

Conduct of this study is justified as it:

1. Assesses a minimal pill count and dosing frequency strategy of co-treatment of HIV and HCV using well tolerated medications with an excellent safety profile and known DDI profile (Complera followed by LPV-SOF). Polypharmacy in the co-infected population remains a significant challenge to therapeutic success.
2. Provides additional safety data for TAF in the HIV-HCV co-infected population.
3. Quantifies adherence and identifies obstacles to full adherence in this population. There is a paucity of data related to DAA adherence in licensing studies.
4. Provides real-world safety and efficacy data to support the public funding for LPV-SOF DAA therapy in HIV-HCV co-infected populations.
5. Provides preliminary data on the immunologic and metabolic consequences of HCV clearance in HIV-HCV co-infection
6. As a pilot study, the information gathered will inform the feasibility of future clinical trials evaluating novel treatment strategies for HIV-HCV co-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected (ELISA with western blot confirmation)
* HCV RNA positive for minimum of 6 months / Genotype 1
* Prescribed cART that may include any Department of Health and Human Services (DHHS) recommended or alternative regimens, which the treating physician considers, is appropriate for their patient. (We anticipate that approximately 60% will be on HIV protease inhibitor-based regimens).
* HIV RNA BLLQ for minimum of 3 months
* Stage 3 or 4 fibrosis
* No evidence of liver decompensation defined as past or current ascites, bleeding varices or hepatic encephalopathy. Prior interferon, ribavirin and/or HCV protease inhibitor exposure will be allowed with the exception of cirrhotic with a past history of null response to interferon-based therapy.
* Ability to remain adherent to medications and study protocol as per investigator opinion
* For female subjects, not pregnant, planning or suspected to be pregnant or breast-feeding
* Willing to use acceptable methods of birth control, as defined in protocol
* Active substance use and/or mental health issues will not be exclusionary assuming other criteria are met. This inclusion will be restricted to those stably housed and engaged in harm reduction strategies. Our intent is to evaluate study participants who are representative of our clinical population and consider 'difficult to cure' compared to populations already evaluated in licensing studies

Exclusion Criteria:

* Concomitant use of drugs with contraindication drug interactions with E/C/F/TAF of SOF-LDV
* History of HIV integrase inhibitors or NRTI resistance mutations
* Platelets <50 x10^9/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Proportion of approached patients who agreed to switch from their current Antiretroviral (ARV) regimen and be screened for this study | 52 weeks
  Number of patients

SECONDARY OUTCOMES:
Proportion of subjects achieving SVR12 | 24 weeks
  HCV RNA at 12 weeks post HCV treatment completion
Proportion of subjects maintaining undetectable HIV RNA levels | 32 weeks
  HIV RNA below detection throughout study period
Proportion of subjects initiating HCV antiviral therapy | 4 weeks
  Number of participants
Proportion of subjects discontinuing study medications due to adverse events | 32 weeks
  Liver enzyme abnormalities

OTHER OUTCOMES:
Measures of fibrosis will be assessed over the duration of the study. | 32 weeks
  Serial Fibroscan assessment at screening, week 12 of Ledipasvir/Sofosbuvir (LDV/SOF) dosing, and 12 weeks after HCV treatment.
Measures of serial cellular immune will be assessed over the duration of the study. | 32 weeks
  CD4 cell counts at Baseline, week 4, week 12, and 12 weeks post treatment
Measures of serial cytokine immune function will be assessed over the duration of the study. | 32 weeks
  Blood will be drawn at each time point for measurement of adipokines (e.g. adiponectin, retinal binding protein 4, interleukin 6, resistin, leptin, visfatin and omentin). (Blood volume: 20 ml).
Measures of metabolic function (cholesterol) will be assessed over the duration of the study | 32 weeks
  Serial measurement of cholesterol at Baseline, week 4, week 12, and 12 weeks post treatment
Measures of metabolic function (glucose) will be assessed over the duration of the study | 32 weeks
  Serial measurement of glucose at Baseline, week 4, week 12, and 12 weeks post treatment
Measures of metabolic function (insulin) will be assessed over the duration of the study | 32 weeks
  Serial measurement of insulin at Baseline, week 4, week 12, and 12 weeks post treatment
Measures of metabolic function (lipokine) will be assessed over the duration of the study | 32 weeks
  Serial measurement of lipokine at Baseline, week 4, week 12, and 12 weeks post treatment
Patient-focused outcome - Quality of life measure will be evaluated | 32 weeks
  EuroQol 5-Dimensional (EQ-5D) questionnaire completed at weeks -4, Baseline, 4, 12 and 12 weeks post treatment to allow for assessment of quality-of-life through quality-adjusted life year (QALY) calculation
Patient-Focused Outcome - Physical Activity will be evaluated | 32 weeks
  International Physical Activity Questionnaire Short-Form (IPAQ-sf) completed at baseline, week 4 and 12 to quantify total physical activity over the past 7 days reported as metabolic equivalent of task (MET) minutes per week across 4 domains: leisure, domestic, work, and transportation-related activities. IPAQ-sf classifies a total combined weekly physical activity score represented as high, moderate, or low activity.
Patient-Focused Outcome - Dietary status will be evaluated | 32 weeks
  Block 2005 Food Frequency Questionnaire (FFQ) completed at baseline, week 12 and 12 weeks post treatment to assess dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Cooper, MD, FRCPC, Principal Investigator — The Ottawa Hospital; Ottawa Hospital Research Institute; Marina Klein, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison ME, Wreghitt T, Palmer CR, Alexander GJ. Evidence for a link between hepatitis C virus infection and diabetes mellitus in a cirrhotic population. J Hepatol. 1994 Dec;21(6):1135-9. doi: 10.1016/s0168-8278(05)80631-2. PMID 7699240
- [Background] Mavrogiannaki A, Karamanos B, Manesis EK, Papatheodoridis GV, Koskinas J, Archimandritis AJ. Prevalence of glucose intolerance in patients with chronic hepatitis B or C: a prospective case-control study. J Viral Hepat. 2009 Jun;16(6):430-6. doi: 10.1111/j.1365-2893.2009.01077.x. Epub 2009 Feb 6. PMID 19200136
- [Background] Grasso A, Malfatti F, De Leo P, Martines H, Fabris P, Toscanini F, Anselmo M, Menardo G. Insulin resistance predicts rapid virological response in non-diabetic, non-cirrhotic genotype 1 HCV patients treated with peginterferon alpha-2b plus ribavirin. J Hepatol. 2009 Dec;51(6):984-90. doi: 10.1016/j.jhep.2009.07.008. Epub 2009 Jul 23. PMID 19695729
- [Background] Poustchi H, Negro F, Hui J, Cua IH, Brandt LR, Kench JG, George J. Insulin resistance and response to therapy in patients infected with chronic hepatitis C virus genotypes 2 and 3. J Hepatol. 2008 Jan;48(1):28-34. doi: 10.1016/j.jhep.2007.07.026. Epub 2007 Oct 1. PMID 17977612
- [Background] Taura N, Ichikawa T, Hamasaki K, Nakao K, Nishimura D, Goto T, Fukuta M, Kawashimo H, Fujimoto M, Kusumoto K, Motoyoshi Y, Shibata H, Abiru N, Yamasaki H, Eguchi K. Association between liver fibrosis and insulin sensitivity in chronic hepatitis C patients. Am J Gastroenterol. 2006 Dec;101(12):2752-9. doi: 10.1111/j.1572-0241.2006.00835.x. Epub 2006 Oct 6. PMID 17026566
- [Background] Hung CH, Wang JH, Hu TH, Chen CH, Chang KC, Yen YH, Kuo YH, Tsai MC, Lu SN, Lee CM. Insulin resistance is associated with hepatocellular carcinoma in chronic hepatitis C infection. World J Gastroenterol. 2010 May 14;16(18):2265-71. doi: 10.3748/wjg.v16.i18.2265. PMID 20458764
- [Background] Baid S, Cosimi AB, Farrell ML, Schoenfeld DA, Feng S, Chung RT, Tolkoff-Rubin N, Pascual M. Posttransplant diabetes mellitus in liver transplant recipients: risk factors, temporal relationship with hepatitis C virus allograft hepatitis, and impact on mortality. Transplantation. 2001 Sep 27;72(6):1066-72. doi: 10.1097/00007890-200109270-00015. PMID 11579302
- [Background] Butt AA, Xiaoqiang W, Budoff M, Leaf D, Kuller LH, Justice AC. Hepatitis C virus infection and the risk of coronary disease. Clin Infect Dis. 2009 Jul 15;49(2):225-32. doi: 10.1086/599371. PMID 19508169
- [Background] Donadon V, Balbi M, Ghersetti M, Grazioli S, Perciaccante A, Della Valentina G, Gardenal R, Dal Mas M, Casarin P, Zanette G, Miranda C. Antidiabetic therapy and increased risk of hepatocellular carcinoma in chronic liver disease. World J Gastroenterol. 2009 May 28;15(20):2506-11. doi: 10.3748/wjg.15.2506. PMID 19469001
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Dai CY, Chuang WL, Ho CK, Hsieh MY, Huang JF, Lee LP, Hou NJ, Lin ZY, Chen SC, Hsieh MY, Wang LY, Tsai JF, Chang WY, Yu ML. Associations between hepatitis C viremia and low serum triglyceride and cholesterol levels: a community-based study. J Hepatol. 2008 Jul;49(1):9-16. doi: 10.1016/j.jhep.2008.03.016. Epub 2008 Apr 22. PMID 18486265
- [Background] Economou M, Milionis H, Filis S, Baltayiannis G, Christou L, Elisaf M, Tsianos E. Baseline cholesterol is associated with the response to antiviral therapy in chronic hepatitis C. J Gastroenterol Hepatol. 2008 Apr;23(4):586-91. doi: 10.1111/j.1440-1746.2007.04911.x. Epub 2007 May 13. PMID 17498221
- [Background] Petit JM, Benichou M, Duvillard L, Jooste V, Bour JB, Minello A, Verges B, Brun JM, Gambert P, Hillon P. Hepatitis C virus-associated hypobetalipoproteinemia is correlated with plasma viral load, steatosis, and liver fibrosis. Am J Gastroenterol. 2003 May;98(5):1150-4. doi: 10.1111/j.1572-0241.2003.07402.x. PMID 12809841
- [Background] Siagris D, Christofidou M, Theocharis GJ, Pagoni N, Papadimitriou C, Lekkou A, Thomopoulos K, Starakis I, Tsamandas AC, Labropoulou-Karatza C. Serum lipid pattern in chronic hepatitis C: histological and virological correlations. J Viral Hepat. 2006 Jan;13(1):56-61. doi: 10.1111/j.1365-2893.2005.00655.x. PMID 16364083
- [Background] Corey KE, Kane E, Munroe C, Barlow LL, Zheng H, Chung RT. Hepatitis C virus infection and its clearance alter circulating lipids: implications for long-term follow-up. Hepatology. 2009 Oct;50(4):1030-7. doi: 10.1002/hep.23219. PMID 19787818
- [Background] Tada S, Saito H, Ebinuma H, Ojiro K, Yamagishi Y, Kumagai N, Inagaki Y, Masuda T, Nishida J, Takahashi M, Nagata H, Hibi T. Treatment of hepatitis C virus with peg-interferon and ribavirin combination therapy significantly affects lipid metabolism. Hepatol Res. 2009 Feb;39(2):195-9. doi: 10.1111/j.1872-034X.2008.00439.x. Epub 2008 Nov 5. PMID 19054155
- [Background] Moucari R, Forestier N, Larrey D, Guyader D, Couzigou P, Benhamou Y, Voitot H, Vidaud M, Seiwert S, Bradford B, Zeuzem S, Marcellin P. Danoprevir, an HCV NS3/4A protease inhibitor, improves insulin sensitivity in patients with genotype 1 chronic hepatitis C. Gut. 2010 Dec;59(12):1694-8. doi: 10.1136/gut.2010.219089. Epub 2010 Sep 21. PMID 20861007
- [Background] Lucidarme D, Foucher J, Le Bail B, Vergniol J, Castera L, Duburque C, Forzy G, Filoche B, Couzigou P, de Ledinghen V. Factors of accuracy of transient elastography (fibroscan) for the diagnosis of liver fibrosis in chronic hepatitis C. Hepatology. 2009 Apr;49(4):1083-9. doi: 10.1002/hep.22748. PMID 19140221
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Hull MW, Rollet K, Moodie EE, Walmsley S, Cox J, Potter M, Cooper C, Pick N, Saeed S, Klein MB; Canadian Co-infection Cohort Study Investigators. Insulin resistance is associated with progression to hepatic fibrosis in a cohort of HIV/hepatitis C virus-coinfected patients. AIDS. 2012 Sep 10;26(14):1789-94. doi: 10.1097/QAD.0b013e32835612ce. PMID 22739388
- [Background] Moreno M, Bataller R. Cytokines and renin-angiotensin system signaling in hepatic fibrosis. Clin Liver Dis. 2008 Nov;12(4):825-52, ix. doi: 10.1016/j.cld.2008.07.013. PMID 18984469
- [Background] Yu JW, Sun LJ, Zhao YH, Kang P, Yan BZ. The effect of metformin on the efficacy of antiviral therapy in patients with genotype 1 chronic hepatitis C and insulin resistance. Int J Infect Dis. 2012 Jun;16(6):e436-41. doi: 10.1016/j.ijid.2012.02.004. Epub 2012 Apr 7. PMID 22486858
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926